CLINICAL TRIAL: NCT00597597
Title: A Phase II Open-Label Trial to Evaluate the Efficacy and Toxicity of Tarceva (Erlotinib) in Women With Metastatic, Hormone Receptor Negative and Her2-Negative Breast Cancer
Brief Title: Phase II Open-Label Trial of Tarceva in Women With Metastatic, Hormone- and HER2-Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough patients enrolled
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ruta Rao, M.D., Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-TAR-721 | L06112402
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; ER and PR hormone receptor negative; HER2/neu negative; EGFR positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label Erlotinib (Experimental): Open label; In this open label study, all enrolled subjects receive active drug, Erlotinib
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — During the treatment period, subjects will receive single agent erlotinib, 150mg/day.
  Other Names: Tarceva

SUMMARY:
The goal of this trial is to determine the activity of erlotinib in a rationally selected population of women with ER-negative, PR-negative, HER2/neu-negative, EGFR-positive breast cancer. If erlotinib is shown to have activity, this could identify a form of targeted therapy for this specific subset of breast cancer patients. In addition, it may identify a subset of breast cancer patients with tumors that overexpress EGFR in whom other EGFR targeted therapies could warrant further testing.

DETAILED DESCRIPTION:
This is a Phase II, open-label, single institution trial of treatment with single agent erlotinib. The purpose of the research is to determine the effects erlotinib has on the breast cancer tumors in women with metastatic hormone receptor negative and HER2-negative breast cancer. The Federal Drug Administration (FDA) has approved erlotinib, also known as Tarceva, for the treatment of locally advanced and metastatic non-small cell lung cancer.

To qualify for the trial, subjects must have histologically confirmed, incurable, locally advanced or metastatic breast cancer that is ER-negative, PR-negative, Her2/neu-negative and EGFR-positive. Subjects must have measurable disease. They must have received less than or equal to 1 chemotherapeutic agent in the metastatic setting. The target accrual is 43 subjects. Initially, 18 subjects will be accrued. If at least 3 subjects are progression-free at 4 months, accrual will continue to a maximum of 43 subjects. Subject eligibility will be evaluated during a screening period of 4 weeks. During the treatment period, subjects will receive single agent erlotinib, 150mg/day. Subjects will receive the first dose of erlotinib on Day 0, within 7 days of registration. Efficacy will be assessed by radiographic tumor assessment or photographic documentation. Safety will be assessed by the recording of adverse events and laboratory test results. Subjects with documented progressive disease will be discontinued from treatment and will be followed for survival information every 2 months until death, lost to follow-up or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Verbal and written informed consent to participate in the study.
2. Women greater than or equal to 18 years of age.
3. Histologically documented metastatic or locally advanced, incurable breast cancer with a tumor block available
4. Less than or equal to 1 prior chemotherapy for metastatic or locally unresectable disease.
5. Prior treatment with anthracycline and taxane chemotherapy, either in the adjuvant or metastatic setting
6. Measurable disease on CT or PET scan or physical exam Disease at a previously irradiated site is considered measurable if there is clear evidence of disease progression following radiation therapy.
7. ER-negative, PR-negative and HER2-neu-negative. Estrogen and progesterone status will be defined by immunohistochemistry. Her2/neu status will be considered negative if the ratio of the number of copies of the Her2/neu gene to the centromeric probe for chromosome 17 is approximately 1. This will be done by FISH (fluorescent in-situ hybridization) testing.
8. EGFR-positive defined as strong membrane staining in greater than 10% of tumor cells by immuno-histochemistry (Dako).
9. Pre- or post-menopausal.
10. ECOG performance status of 0 - 2.
11. Life expectancy of greater than or equal to 3 months.
12. Use of barrier contraceptive methods in women of childbearing potential.
13. Ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. Pleural effusions or blastic bone lesions as the only manifestations of the current metastatic breast cancer.
2. Other primary malignancies within 5 years except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer.
3. Symptomatic or untreated brain metastases. Subjects are eligible if they are neurologically stable after treatment for brain metastases and have been off steroids for greater than or equal to 4 weeks.
4. Radiotherapy, immunotherapy, hormonal therapy or chemotherapy within 21 days prior to registration.
5. Prior treatment with an agent that targets the EGFR or the EGFR-specific tyrosine kinase activity.
6. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 0, or serious cardiac arrhythmias requiring medication.
7. Major surgery, biopsy of a parenchymal organ, or significant traumatic injury occurring within 21 days prior to Day 0.
8. History of other diseases, metabolic dysfunction, physical examinations findings, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications.
9. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
10. Pregnancy or lactation. A negative serum or urine pregnancy test is required for women of child-bearing potential during screening and within 7 - 10 days of Day 1 of Cycle 1 of erlotinib (Tarcevo®)administration. Men and premenopausal women of child bearing potential will follow an approved, medically accepted birth control regimen while taking erlotinib and for 30 days following the last dose of study drug.
11. Active infection requiring parenteral antibiotics.
12. Any of the following abnormal baseline hematologic values:

    * Granulocyte count less than or equal to 1500/μL
    * Platelet count less than or equal to 100,000/μL
    * Hemoglobin less than or equal to 9g/dl (transfusion permitted)
13. Any of the following abnormal baseline liver function tests:

    * Serum bilirubin greater than or equal to 1.5x upper limit of normal (ULN)
    * Serum ALT and AST greater than or equal to 2.5x ULN (greater than 5x ULN if due to liver metastases)
    * Alkaline phosphatase greater than or equal to 2.5x ULN (greater than 4x ULN if due to liver or bone metastases)
14. Other baseline laboratory values:

    * Serum creatinine greater than or equal to 1.5x ULN or creatinine clearance less than or equal to 60mL/min
    * Uncontrolled hypercalcemia (greater than 11.5mg/dL)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruta D Rao, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center Division of Hematology/Oncology, Chicago, Illinois, United States

REFERENCES:
- [Result] J Clin Oncol 29, 2011 (suppl 27; abstr 296)

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: 150mg/Day: Erlotinib: 150mg/day.
Period: Overall Study
Arm/Group | Erlotinib: 150mg/Day
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- A Phase II Open-Label Clinical Trial to Evaluate the Efficacy: Open label; all subjects receive active drug, Erlotinib
  Erlotinib: During the treatment period, subjects will receive single agent erlotinib, 150mg/day.
  All patients receive the study drug, erlotinib, at the dose of 150 mg/day
  Patients were eligible if they had locally recurrent or metastatic breast cancer that was triple negative and positive for EGFR. EGFR positivity was defined as staining in >10% of tumor cells by immunohistochemistry (Dako). Patients required measurable disease on imaging or physical examination, prior treatment with anthracycline and taxane (either in adjuvant or metastatic setting) and ≤1 prior chemotherapy in the metastatic setting. Patients received erlotinib 150mg daily.
Arm/Group | A Phase II Open-Label Clinical Trial to Evaluate the Efficacy
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [40 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is Progression Free Survival.
Description: From the Day of Initial Treatment (Day 0) Until Documented Disease Progression or Death.
Time Frame: From the Day of Initial Treatment (Day 0) Until Documented Disease Progression or Death, whichever came first, assessed up to 6 months.
Measure: Median (Standard Deviation); unit: years
Groups:
- A Phase II Open-Label Clinical Trial to Evaluate the Efficacy: Open label; all subjects receive active drug, Erlotinib
  Erlotinib: During the treatment period, subjects will receive single agent erlotinib, 150mg/day.
Arm/Group | A Phase II Open-Label Clinical Trial to Evaluate the Efficacy
Number analyzed (Participants) | 11
years | 0.08 (1.2)

2. Secondary Outcome: Overall Response Rate, Consisting of Complete and Partial Responses According to RECIST Criteria
Description: Overall response rate, consisting of complete and partial responses according to RECIST criteria "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: every 8 weeks, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib: 150mg/Day
Number analyzed (Participants) | 11
Participants | 0

3. Secondary Outcome: Clinical Benefit, Consisting of Complete and Partial Responses, and Stable Disease for Six Months
Description: We measured the clinical benefit, consisting of complete and partial responses, and stable disease for six months
Time Frame: very 8 weeks, up to 6 months
Measure: Number; unit: participants
Arm/Group | Erlotinib: 150mg/Day
Number analyzed (Participants) | 10
participants | 2

4. Secondary Outcome: Duration of Objective Response
Description: Objective response is defined as complete or partial response
Time Frame: every 8 weeks, up to 6 months
Population: 0 patients were observed to have an objective response
Arm/Group | Erlotinib: 150mg/Day
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety of Erlotinib
Description: Number of Participants With Adverse Events
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Erlotinib: 150mg/Day
Number analyzed (Participants) | 11
participants | 2

6. Secondary Outcome: Number of Participants With Rash
Description: We evaluated the number of Participants with Rash
Time Frame: every 8 weeks, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib: 150mg/Day
Number analyzed (Participants) | 11
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | A Phase II Open-Label Clinical Trial to Evaluate the Efficacy
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Phase II Open-Label Clinical Trial to Evaluate the Efficacy (N=11)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
diarrhea (Gastrointestinal disorders) | 2 (2) — Grade 1
nausea (Gastrointestinal disorders) | 1 (1) — Grade 1
weight loss (General disorders) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No